CLINICAL TRIAL: NCT05917808
Title: A Food Product for Glucose Management in Gestational Diabetes Mellitus - a Pilot Study
Brief Title: Food Product for Management of Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stoffwechselzentrum Rhein - Pfalz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMP2301
Record Dates: First submitted 2023-05-25; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes; Glucose Tolerance Impaired in Pregnancy; Glucose Tolerance Impaired; Pregnancy Related; Insulin Sensitivity/Resistance
Keywords: Wholegrain; Dietary Intervention; Gestational Diabetes; Impaired Glucose Tolerance; Insulin Sensitivity/Resistance
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: single-center, non-randomized, open, pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Only study arm in the study. Participants consume a ready-to-eat wholegrain porridge on two consecutive evenings and repeat OGTT
  Interventions: Other: Ready-to-eat wholegrain porridge

INTERVENTIONS:
Other: Ready-to-eat wholegrain porridge — A ready-to-eat wholegrain porridget will be consumed shortly after a diagnostic OGTT on two consecutive evenings, the OGTT will then be repeated

SUMMARY:
The goal of this pilot open pre-post clinical trial is to test effects of a wholegrain product in patients with newly diagnosed gestational diabetes. The main question it aims to answer is:

Does the wholegrain product improve glucose tolerance and insulin sensitivity during a 75 g oral glucose tolerance test (OGTT).

Participants will consume product on two consecutive evenings shortly after the first OGTT and will then perform a second OGTT. Researchers will compare the results of the first and second OGTT to see if glucose tolerance improved after consumption of the test product.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological fasting glucose or OGTT according to WHO-criteria for the diagnosis of gestational diabetes (see Table 1).
2. Agree to maintain consistent dietary habits and physical activity levels for the duration of the study.
3. Willingness to complete questionnaires and follow instructions associated with the study and to perform another OGTT at the clinic in a second visit.
4. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Type 2 diabetes prior to pregnancy
2. Psychiatric Disease
3. Acute Infections
4. Alcohol or drug abuse
5. Acute diverticulitis
6. Malignant tumors or hematologic disorders
7. Heart failure stages III-IV according to New York Heart Association (NYHA)
8. Acute coronary syndrome
9. Chronic kidney disease > Stage 3 (Kidney Disease Outcomes Quality Initiative - KDOQI)
10. Celiac disease
11. Diagnosed Inflammatory bowel diseases (mainly Crohn´s, Ulcerative colitis)
12. Allergy to ingredients included in the investigational product.
13. Use of antibiotics within 2 weeks of enrollment
14. Use of probiotics within 2 weeks of enrollment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women with gestational diabetes
Enrollment: 25 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 2 hour glucose in OGTT | 3-7 working days
  Change of the 2 hour glucose value in an oral glucose tolerance test

SECONDARY OUTCOMES:
Change of the fasting glucose values | 3-7 working days
  Change in in fasting plasma glucose
Change in 1h glucose in OGTT | 3-7 working days
  Change of the 1h glucose value in an oral glucose tolerance test from the first to the second OGTT
Number of values changing from diabetic to non-diabetic values per patient | 3-7 working days
  Number of values changing from above the diabetic threshold to below diabetic threshold per patient in the cohort according to World Health Organization (WHO) definitions
Number of individuals converting from diabetic to non-diabetic OGTT / fasting glucose | 3-7 working days
  Number of individuals converting from diabetic to non-diabetic OGTT / fasting glucose according to WHO criteria
Change in plasma insulin fasting | 3-7 working days
  Change in plasma insulin fasting between 1st and second OGTT
Change in plasma insulin 1 hour during OGTT | 3-7 working days
  Change in plasma insulin 1 hour during OGTT between 1st and second OGTT
Change in plasma insulin 2 hour during OGTT | 3-7 working days
  Change in plasma insulin 2 hour during OGTT between 1st and second OGTT
Change in homeostasis model assessment (HOMA) Index between 1st and second OGTT | 3-7 working days
  Change in HOMA Index between 1st and second OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Stoffwechselzentrum Rhein-Pfalz, Mannheim, Baden-Wurttemberg, Germany